CLINICAL TRIAL: NCT02661425
Title: Retrospective Study of Irritable Bowel Syndrome With Diarrhea (IBS-D) Patients Previously Receiving Serum-derived Bovine Serum Immunoglobulin (SBI)
Brief Title: Retrospective Study of IBS-D Patients Previously Receiving SBI
Status: Completed | Type: Observational
Sponsor: Entera Health, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EH MA 1010
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Diarrhoea Predominant Irritable Bowel Syndrome
Keywords: IBS-D; IBS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard of Care
- EnteraGam
  Interventions: Other: EnteraGam

INTERVENTIONS:
Other: EnteraGam — Serum-derived bovine immunoglobulin/protein isolate (SBI) is the nutritional ingredient in EnteraGam. SBI contains a minimum of 50% immunoglobulin. The protein isolate is a light-colored powder. Each packet contains SBI (5.0 g) and the following inactive ingredients: dextrose (5.0 g) and a trace amount of sunflower lecithin.
  Other Names: Serum-Derived Bovine Immunoglobulin/Protein Isolate
  Groups: EnteraGam

SUMMARY:
This is a retrospective study designed to gather outcomes data from existing medical charts from patients who have taken EnteraGam for management of their IBS-D for at least eight weeks. Data from two study periods will be collected: (1) the time during which the Standard of Care (SOC) therapy (i.e., prescribed or over-the-counter as well as FDA-approved or non-approved agents) that is used immediately prior to prescribing EnteraGam; and (2) the time during which EnteraGam is used as therapy.

DETAILED DESCRIPTION:
* The first collection of information (Visit 1 - Chart Report Form) will be for the visit at which the SOC therapy, utilized immediately before the introduction of EnteraGam, was initiated. This data point will serve as the baseline for that SOC therapy.
* The second collection of information (Visit 2 - Chart Report Form) will be for the visit at which the original prescription for EnteraGam was written and the patient was instructed to begin the therapy. Captured data will consist of information contained in the patient's chart for a minimum of eight weeks and a maximum of 12 weeks prior to initiation of EnteraGam therapy. This data point will serve as the baseline for initiation of EnteraGam therapy.
* The third collection point (Visit 3 - Chart Report Form) will be at the next patient visit to the clinic - provided that visit is a minimum of eight weeks following initiation of EnteraGam therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age at the initiation of EnteraGam therapy.
* Patient has been previously diagnosed with IBS-D by the physician and has undergone at least one course of SOC treatment prior to receiving EnteraGam.
* Patient has completed a minimum of eight weeks of EnteraGam therapy for his / her IBS-D.
* There is recorded information regarding patient response to SOC or EnteraGam for stool frequency/consistency and abdominal pain

Exclusion Criteria:

* Patient has not taken EnteraGam for a minimum of eight weeks or has not used the product according to the directions provided by the prescribing physician.
* Patient has not consented to the use of their clinical data in this retrospective clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have failed on Standard of Care and then taken EnteraGam for management of their IBS-D for at least eight weeks.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Improvement in the combined score for stool frequency/consistency and abdominal pain intensity during the time that the patient is receiving EnteraGam. | minimum of 8 weeks
  Data collected from existing medical charts

SECONDARY OUTCOMES:
Improvement in stool frequency | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in stool consistency | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in abdominal pain intensity | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in urgency | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in flatulence | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in fecal incontinence | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in bloating | minimum of 8 weeks
  Data collected from existing medical charts
Improvement in fatigue | minimum of 8 weeks
  Data collected from existing medical charts

CONTACTS AND LOCATIONS:
Overall Officials: Larry Good, MD, Principal Investigator — South Nassau Communities Hospital
Locations (16):
- United States (16):
  - Greenwich, Connecticut
  - Hamdon, Connecticut
  - Coral Springs, Florida
  - Maitland, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Smyrna, Georgia
  - Columbia, Maryland
  - St Louis, Missouri
  - Lynbrook, New York
  - New York, New York
  - Kingsport, Tennessee
  - Knoxville, Tennessee
  - Morristown, Tennessee
  - Bedford, Texas

IPD SHARING:
Plan to Share IPD: No